CLINICAL TRIAL: NCT06736093
Title: Effect of Preoperative Vitamin D Supplementation in Liver Transplant Recipients With Vitamin D Deficiency on Post Transplant Outcomes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: ILBS-CLDVitaminD-2024
Record Dates: First submitted 2024-11-24; First posted 2024-12-16 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-01

CONDITIONS: Post Liver Transplant Infection
MeSH Terms: interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Vitamin D Supplementation Arm (Active Comparator)
  Interventions: Drug: Vitamin D3
- Placebo Arm (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Vitamin D3 — Vitamin D3 60,000 IU given once weekly Pre Liver Transplant atleast for 6 weeks
  Arms: Vitamin D Supplementation Arm
Drug: Placebo — Placebo capsules once weekly for atleast 6 weeks pre liver transplant
  Arms: Placebo Arm

SUMMARY:
Liver transplantation (LT) remains the ultimate option to cure intractable end stage liver disease. Vitamin D deficiency is very common in these subsets of patients. Vitamin D is involved in calcium metabolism and bone mineralization, regulation of cytokines, immunomodulation, cellular proliferation and differentiation. Its deficiency can lead to immune dysregulation, and is associated with the development of viral and bacterial infections, cardiovascular and autoimmune diseases, and several types of cancer. To the best of our knowledge, there are no randomized studies which analyze the effect of Vitamin D supplementation preoperatively on post Liver Transplant outcomes. This double blinded placebo-controlled randomized study aims to analyze the effect of preoperative supplementation of Vitamin D in patients with Vitamin D deficiency on post liver transplant outcomes. All eligible adult patients with Chronic Liver Disease and Vitamin D deficiency undergoing Liver Transplant during the study period will be included in the study and randomized into two groups. One group will receive Oral Vitamin D3 - 60000 IU - once a week pre Liver Transplant for a minimum of 6 weeks and the other will receive placebo once a week for a minimum of 6 weeks in addition to 3 months Vitamin D supplementation post Liver Transplant in both arms.

All Liver Transplant Recipients with Vitamin D deficiency will be screened in the pre-operative period in the outpatient department. Pre-operative, intra-operative and post-operative data will be collected from medical records, electronic hospital information system (HIS) and radiological images collected from the hospital Picture archiving and communication system(PACS). The enrolled subjects will be followed up till for a period of 3 months after the Liver Transplant and the post transplant bacterial infection rates will be compared between the two groups along with other parameters.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients >18 yrs with Cirrhosis of Liver and Vitamin D deficiency ( defined as levels < 30 ng/ml) undergoing Liver Transplant.

Exclusion Criteria:

* Negative consent Pediatric patients Infection at the time of Liver Transplant Acute Liver Failure Deceased Donor Liver Transplant Patients undergoing Re Liver Transplant Patients already receiving Vitamin D supplements. Patients with Hypoparathyroidism/ Hyperparathyroidism H/o other Solid Organ Transplantation Patients needing urgent Liver transplant before 6 weeks of Vitamin D Supplementation.

Patients with Vitamin D levels < 10 ng/ml Patients with Osteoporosis ( DEXA BMD T Score <-2.5)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2025-01-10 (Actual); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
To compare the Post Liver Transplant bacterial infection rates in the first 3 months between the two arms. | 3 months post Liver Transplant

SECONDARY OUTCOMES:
To compare the Acute Graft Rejection rates between the two arms within 3 months post liver transplant | 3 months
To compare the Sepsis (Bacterial and Fungal) and septic shock rate between the two arms within 3 months post liver transplant | 3 months
To compare the Serum Vitamin D3 levels between the two arms at 3 months post liver transplant. | 3 months
To compare the Bone mineral Density (T score) between the two arms at 3 months post liver transplant. | 3 months
To compare Bone formation markers-Osteocalcin (OC),Osteoprotegerin (OPG) and bone resorption markers -carboxyl-terminal telopeptide of type 1 collagen (CTX-1), Bone-specific Alkaline Phosphatase (BALP) between the two arms 3 months post liver transplant. | 3 months
To compare the Overall Survival between the two arms 3 months post liver transplant. | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Nihar Mohapatra, MS, MCh, Study Director — Institute of Liver and Biliary Sciences, New Delhi, India; Sridhar L, MS, Principal Investigator — Institute of Liver and Biliary Sciences, New Delhi, India
Locations (1):
- Institute of Liver and Biliary Sciences, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: No